CLINICAL TRIAL: NCT05932381
Title: Effect Of Complete Decongestive Therapy On Carpal Tunnel Syndrome Post Upper Limb Lymphedema
Acronym: CDT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Abd Elmohsen Ali, principle investigator Sara Abd Elmohsen Ali, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003738
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Lymphedema
Keywords: complete decongestive therapy; carpal tunnel syndrome; upper limb lymphedema
MeSH Terms: conditions — Lymphedema; Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: complete decongestive therapy and routine medical treatment
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complete decongestive therapy (Experimental): the patients will receive complete decongestive therapy twice a week for ten weeks
  Interventions: Other: Complete decongestive therapy; Other: Medical treatment
- medical treatment (Active Comparator): the patients will receive routine medical treatment for ten weeks
  Interventions: Other: Medical treatment

INTERVENTIONS:
Other: Complete decongestive therapy — the patients will receive Complete decongestive therapy in the form of intermittent pneumatic compression, Exercising, bandaging, and manual lymphatic drainage with Pressures of 50, 80, and 120 mmHg and timing 5, 20, and 50 secs
  Arms: Complete decongestive therapy
Other: Medical treatment — the patients will receive routine medical treatment

SUMMARY:
this study will be conducted to investigate the therapeutic effect of complete decongestive therapy on carpal tunnel syndrome post-upper limb lymphedema.

DETAILED DESCRIPTION:
lymphedema is a chronic condition characterized by lymphatic vessel ectasia and valve dysfunction, followed by the reflux of lymphatic fluid into the interstitial space. Lymph stasis may lead to a chronic inflammatory process, resulting in adipose tissue differentiation and fibro adipose tissue deposition. One consequence of post-mastectomy lymphedema may be the development of nerve entrapments. One example is median nerve entrapment in the carpal canal, or carpal tunnel syndrome (CTS). many studies assessed the relationship of CTS as a risk factor for developing lymphedema, other studies stated the possibility of lymphedema as a potential contributor to CTS development. Complex decongestive treatment of breast cancer-related lymphoedema is an accepted strategy and is considered as an international standard for treatment. A previous review concluded that complex decongestive therapy has a positive impact on the volume of arm and quality of life in different stages of lymphedema.sixty females will be allocated randomly to two groups; first one will receive decongestive therapy and the second one will receive the routine medical treatment for ten weeks

ELIGIBILITY:
Inclusion Criteria:

* Age will range between 20- 40 years.
* Only females will participate in the study.
* All patients have carpal tunnel syndrome post upper limb lymphedema.

Exclusion Criteria:

* Diabetes mellitus.
* Individuals with cardiopulmonary conditions.
* Individuals undergoing radiation therapy or chemotherapy.
* Hepatic or pancreatic diseases.
* Sensory impairment.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-05 (Estimated); Primary Completion 2023-10-05 (Estimated); Study Completion 2023-10-05 (Estimated)

PRIMARY OUTCOMES:
hand strength | up to ten weeks
  hand held dynamometer will be used for measuring the hand strength
median nerve conduction velocity | up to ten weeks
  median nerve conduction velocity will be measured by electromyography device

SECONDARY OUTCOMES:
pain intensity | up to ten weeks
  Visual analogue scale which is 100 mm horizontal line will be used for measuring pain intensity. the scale has no pain on the left side and worst pain on the right side